CLINICAL TRIAL: NCT06542952
Title: Statistical Analysis of Prevalence, Incidence, Comorbidities and Medical Expense in Epileptic Children in Taiwan Based on National Health Research Insurance Database
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Professor, National Taiwan University Hospital
Other Study IDs: 201802028RINB
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Neurologic Disorder; Seizure Disorder
MeSH Terms: conditions — Nervous System Diseases; Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: seizure — epileptic children

SUMMARY:
Epilepsy is a common disease in pediatric neurology. In recent years, due to the promotion of Taiwan's health insurance and the advancement of related medical treatments and anti-epileptic drugs, the prevalence, incidence, and related comorbidities of childhood epilepsy in Taiwan are expected, as well as the number of epilepsy patients in different regions or different age groups. and medical costs may change. This study aims to collect data from the National Health Insurance Database through the National Institutes of Health, review relevant data on childhood epilepsy patients from 2001 to 2013, and analyze trends to discuss the impact of universal health insurance and medical progress on childhood epilepsy patients. Impact.

ELIGIBILITY:
Inclusion Criteria:

1. Targets aged 0~19 (<=19) in the home country
2. Diagnosis code includes ICD9: 345.XX, ACODE:A225 (including outpatient and inpatient)
3. Between 2001 and 2013, those who had seen a doctor three times in a row with epilepsy diagnosis codes and used anti-epileptic drugs

Exclusion Criteria:

* Exclude those who sought medical treatment for epilepsy from 2001 to 2013, but the number of medical visits (outpatient + hospitalization) <3 times, and exclude those who did not take medication from 2001 to 2013.

Ages: 0 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients suffering from epilepsy
Sampling Method: Probability Sample
Enrollment: 169026 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Statistical Analysis of prevalence, incidence, comorbidities and medical expense medical expense in epileptic children in Taiwan based | 2001-2013
  in epileptic children in Taiwan based

CONTACTS AND LOCATIONS:
Overall Officials: Mei Lan Liou, master, Study Director — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Tainan
  - Department of Pediatrics, National Taiwan University Hospital, Taipei